CLINICAL TRIAL: NCT04359368
Title: Characteristics of Patients With Hypersensitivity Reactions to Intravenous Iron Infusions - a Retrospective Study
Brief Title: Characteristics of Patients With Hypersensitivity Reactions to Intravenous Iron Infusions
Status: Completed | Type: Observational
Sponsor: University Hospital, Basel, Switzerland (Other)
Responsible Party: Sponsor
Other Study IDs: 2019-01266;sp20Steveling3
Record Dates: First submitted 2020-04-21; First posted 2020-04-24 (Actual); Last update posted 2020-04-24 (Actual); Status verified 2020-04

CONDITIONS: Iron-deficiency; Hypersensitivity Reactions
Keywords: complement activation-related pseudoallergy (CARPA); Hypersensitivity reactions (HSR); iron-deficiency; non dextran iron preparations (NDIPs); anemia
MeSH Terms: conditions — Anemia, Iron-Deficiency; Hypersensitivity; Anemia

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- patients with hypersensitivity reactions to NDIPs: Patients with previous hypersensitivity reaction grades I-IV to intravenous ferric carboxymaltose (Ferinject) or to iron sucrose (Venofer)
  Interventions: Other: collection of patient data

INTERVENTIONS:
Other: collection of patient data — Data collection (history, clinical presentation, medication, complications, laboratory testing) will be performed from patient records stored in the protected electronic patient system ISMed (Integrated System for Medical Diagnostic) of patients with HSRs to NDIPs.

SUMMARY:
This study aims to evaluate characteristics of patients with previous hypersensitivity reaction grades I-IV to intravenous ferric carboxymaltose (Ferinject) or to iron sucrose (Venofer) including age, atopy status, previous allergic reactions, previous medical history, current medications and co-morbidities. Furthermore, symptoms on reaction such as severity grade of reaction will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Participants from 16 years of age and older with previous hypersensitivity reaction grades I-IV to intravenous ferric carboxymaltose (Ferinject) or to iron sucrose (Venofer).

Exclusion Criteria:

* No previous hypersensitivity reaction to iron preparations or reactions to oral iron preparations.
* If a rejection to use patient data is documented in patient records, the patient will be excluded from analysis.

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Participants from 16 years of age and older with previous hypersensitivity reaction grades I-IV to intravenous ferric carboxymaltose (Ferinject) or to iron sucrose (Venofer).
Sampling Method: Probability Sample
Enrollment: 42 (Actual)
Dates: Start 2019-09-01 (Actual); Primary Completion 2019-10-31 (Actual); Study Completion 2019-10-31 (Actual)

PRIMARY OUTCOMES:
previous medical history | Baseline; Patients with HSRs to NDIPs that were treated at the University Hospital Basel between the 16th of January 2018 and the 24th of October 2019
  Data collection (medical history) will be performed from patient records stored in the protected electronic patient system ISMed (Integrated System for Medical Diagnostic) of patients with HSRs to NDIPs
Family history | Baseline; Patients with HSRs to NDIPs that were treated at the University Hospital Basel between the 16th of January 2018 and the 24th of October 2019
  Data collection (Family history) will be performed from patient records stored in the protected electronic patient system ISMed (Integrated System for Medical Diagnostic) of patients with HSRs to NDIPs
assessment of hypersensitivity reactions | Baseline; Patients with HSRs to NDIPs that were treated at the University Hospital Basel between the 16th of January 2018 and the 24th of October 2019
  assessment of hypersensitivity reactions (grade I-IV) to Ferinject or Venofer
preparation used | Baseline; Patients with HSRs to NDIPs that were treated at the University Hospital Basel between the 16th of January 2018 and the 24th of October 2019
  which preparation was used for Treatment ( iron sucrose (Venofer) or ferric carboxymaltose (Ferinject)
co-medication | Baseline; Patients with HSRs to NDIPs that were treated at the University Hospital Basel between the 16th of January 2018 and the 24th of October 2019
  which co-medication was used

CONTACTS AND LOCATIONS:
Overall Officials: Esther Steveling-Klein, Dr. med, Principal Investigator — Allergology, University Hospital Basel
Locations (1):
- University Hospital Basel, Basel, Switzerland